CLINICAL TRIAL: NCT06107621
Title: Internet-based Cognitive Behavioral Therapy for Gambling Disorder and and Comorbidities - a Pilot Study
Brief Title: iCBT for GD and Comorbidities - a Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Deakin University (Other)
Responsible Party: Principal Investigator, Olof Molander, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2023-01074-01
Record Dates: First submitted 2023-08-30; First posted 2023-10-30 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Gambling Disorder; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-based iCBT targeting Gambling Disorder and comorbidities (Experimental): An 8 module internet-based iCBT program targeting Gambling Disorder and comorbidities, administered with treatment support.
  Interventions: Behavioral: iCBT for Gambling Disorder and psychiatric comorbidities

INTERVENTIONS:
Behavioral: iCBT for Gambling Disorder and psychiatric comorbidities — The iCBT, is based on the gambling pathways model. As a clinical conceptualization, the treatment build on loss of control, but also include additional interventions (e.g., emotion regulation and impulse control) targeting the etiological co-morbidity factors in the pathways model for emotionally vulnerable and impulsive gamblers (pathways subtypes 2 and 3).

SUMMARY:
The study is a pilot study (Total N=30), with at pre, weekly during treatment, post and at three-month follow-up.

DETAILED DESCRIPTION:
Recruitment will be done through online advertisement via social media and gambling-related websites. Participants will self-referred to the study via a study dedicated website (www.spelstudien.se). Login to a treatment platform will be verified using double authentication (detailed description of the online platform is provided in the application to the Swedish Ethical Review Authority). Written information about the study will be provided on the web page. Consent will be done online, with the possibility for participants to download study information and consent. Consenting participants will start a screening procedure. After screening, participants will be contacted for a telephone assessment with a clinical psychologist. During this interview, participants will be assessed for GD with a diagnostic interview, as well as the inclusion criteria for utilization of "Spelpaus".

If meeting criteria for the study, participants will be referred to the baseline/ pre-measures - which will start with an additional informed consent for the treatment phase and the iCBT. Inclusion will be done after the completion of the informed consent and baseline/pre-measures. After that, participant will get access to the iCBT.

ELIGIBILITY:
Inclusion Criteria:

* Screen positive for GD, as measured with the Gambling Disorder Identification Test (total score ≥20 GDIT).
* Fulfilling GD, assessed according to the Structured Clinical Interview for Gambling Disorder (SCI-GD).
* Utilization of "Spelpaus" (3 months from treatment start).
* ≥18 years of age.
* Able to provide digital informed consent.
* Classified within pathways 2 or 3, as measured with the Gambling pathways Questionnaire (GPQ).
* Screen positive for at least one common mental diagnosis in addition to GD, assessed according to the Web Screening Questionnaire (WSQ).

Exclusion Criteria:

* Other ongoing psychological treatment for GD.
* Severe depression, screened according to the Montgomery Åsberg Depression Rating Scale (total score >34 MADRS-S).
* Suicidality, screening of ≥4 points on item 9 of the MADRS-S

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The Gambling Symptom Assessment Scale | Six months after treatment cessation
  Primary outcome will be gambling symptoms, measured with the the Gambling Symptom Assessment Scale. Minimum score is 0 and maximum score is 48, with higher scores indicated higher frequency of gambling symptoms.

SECONDARY OUTCOMES:
The TimeLine Followback for gambling | Six months after treatment cessation
  Gambling behavior (days per week gambled) will be measured with a self-report item adapted from the TimeLine Followback for gambling.
The Generalized Anxiety Disorder 7-itemscale | Six months after treatment cessation
  Anxiety symptoms will be measured by the Generalized Anxiety Disorder 7-itemscale.
The Patient Health Questionnaire | Six months after treatment cessation
  Depressive symptoms will be measured with the The Patient Health Questionnaire.
The Alcohol Use Disorders Identification Test | Six months after treatment cessation
  Alcohol problems will be measured with the Alcohol Use Disorders Identification Test.
The Drug Use Disorders Identification Test | Six months after treatment cessation
  Drug problems will be measured with the Drug Use Disorders Identification Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for psychiatry research, Stockholm, Sweden